CLINICAL TRIAL: NCT05873257
Title: Investigation of the Clinical Performance of Biatain Fiber Ag on Venous Leg Ulcer
Brief Title: Investigation of the Clinical Performance of Biatain Fiber Ag on Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP358
Record Dates: First submitted 2023-05-01; First posted 2023-05-24 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Venous Leg Ulcer
Keywords: wound healing
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: non-comparative, one-armed, open-labelled, multi-centre study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- main arm (Other): Non comparative - One armed - open labelled Intervention - subjects will wear the test dressing in a four weeks period with planned dressing changes once pr. week.
  Interventions: Device: Biatain Fiber Ag applied to participants

INTERVENTIONS:
Device: Biatain Fiber Ag applied to participants — Intervention involving a wound gelling fiber dressing with silver

SUMMARY:
The goal of this study is to test a new gelling fiber wound dressing with silver on patients with a venous leg ulcer

Participants will be asked to wear the test dressing in a four weeks period (+/- 2 days) consisting of 6 study visits, and will have the dressing changed once pr. week at the research facility. The wound will be cleaned, assessed and photos will be uploaded to a digital software system.

DETAILED DESCRIPTION:
: The clinical investigation is a non-comparative, one-armed, open-labelled, multi-centre study

The test product, Biatain Fiber Ag is a non-CE-marked gelling fiber wound dressing, containing silver. The product is intended for moist wound healing and exudate management of moderate to high exuding wounds.

The overall purpose of this investigation is to obtain clinical data supporting effectiveness of Biatain Fiber Ag to obtain the CE-mark in EU.

The total study duration for the subject will be approximately four weeks, consisting of a four-week test period and 6 study visits (V0/V1, V2, V3, V4 and V5). V5 will also terminate the 4-week study period.

The primary endpoint is Mean area wound reduction. The endpoint is used to evaluate clinical performance in terms of relative wound area reduction as an indication of total wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed informed consent
2. Is 18 years or above
3. Is capable of following study procedure (assessed by the investigator).
4. Has a venous leg ulcer that has failed to progress along the expected wound healing trajectory within 4 weeks
5. The shape of the wound should be possible to fit under a 10x10 cm dressing
6. The shape and location of the wound should be suitable for photo capture (assessed by the investigator).
7. Has at least three of five pre-defined clinical signs of infection; pain between two dressing changes, peri-ulcer skin erythema/inflammation, oedema, malodour, or heavy exudate (assessed by the investigator).
8. Has a wound that has medium to high level of exudate (assessed by the investigator).
9. Has an ankle to brachial pressure index (ABPI) of 0.8 -1.3
10. Agrees to wear compression therapy daily in combination with the test dressing
11. Is suitable to use the test product for wound treatment (assessed by the investigator).

Exclusion Criteria:

1. Is pregnant/breastfeeding
2. Wound is older than 12 months
3. Wound with exposed tendons or bones or has fistulas
4. Wound which is undermined or tunneling
5. Is currently receiving or has within the past 60 days received radio- and/or chemotherapy (low doses radio- and/or chemotherapy is allowed for other indications than cancer if assessed by investigator not to influence study wound area)
6. Known history of skin sensitivity to any components of the treatment dressings
7. Intake of antibiotics within one week before the start of the enrolment
8. Participation in any other clinical studies that can compromise this study treatment (assessed by the investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria Healthcare NHS foundation trust, Ashington, Northumbria, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Arm: Non comparative - One armed - open labelled Intervention - subjects will wear the test dressing in a four weeks period with planned dressing changes at least once per week.
  Biatain Fiber Ag applied to participants: Intervention involving a wound gelling fiber dressing with silver
Period: Overall Study
Arm/Group | Main Arm
Started (Safety population/Intention-to-Treat population) | 50
Completed | 45
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Main Arm
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 40
Age, Continuous [Mean (Full Range); unit: years] | 75.4 [21 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50
Wound area [Mean (Full Range); unit: cm2] | 12.3 [1 to 66]
Wound age [Mean (Full Range); unit: weeks] | 22.4 [5 to 52]
Signs of infection in the wound [Number; unit: participants] | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Relative Wound Area Reduction as Indication of Total Wound Healing
Description: Wound area will be measured by obtaining photos of the wounds and measure these afterwards. A planimetric software will be used where the wound is photographed with a ruler of known dimensions placed at the skin near the wound edge and the image is transferred to a computer and opened in the planimetric software. The ruler is used for calibration of linear dimensions at the image. Once the wound border is manually traced with a computer mouse the area of wound is calculated and displayed.
Time Frame: 4 weeks
Population: The primary analysis was based on subjects exposed to investigational device and with reliable baseline assessment of wound area. One subject was omitted (entire wound not captured on photo at baseline). The last observation 'on-treatment' was used in the analysis.
  The sensitivity analysis was conservatively based on the entire ITT population also including a subject with an unreliable wound area assessment at baseline. The analysis was performed as the primary analysis.
Measure: Mean (95% Confidence Interval); unit: relative wound area reduction (%)
Arm/Group | Main Arm
Number analyzed (Participants) | 50
relative wound area reduction (%)
  Primary analysis: number analyzed (Participants) | 49
  Primary analysis | 46.3 [36.5 to 56.2]
  Sensitivity analysis | 43.9 [33.1 to 54.7]

ADVERSE EVENTS:
Time Frame: 4 weeks (+/- 2 days)
Groups:
- Main Arm: Non comparative - One armed - open labelled Intervention - subjects will wear the test dressing in a four weeks period with planned dressing changes once per week.
  Biatain Fiber Ag applied to participants: Intervention involving a wound gelling fiber dressing with silver
Arm/Group | Main Arm
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 8/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Arm (N=50)
Hospitalised with pulmonary oedema (Cardiac disorders) | 1 (1) — Not related to investigational device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Arm (N=50)
Antibiotics prescribed for study wound (Infections and infestations) | 5 (5) — Not related to investigational device
Cellulitis (right hand) (Infections and infestations) | 1 (1) — Not related to investigational device
Increased severe pain at wound site (General disorders) | 1 (1) — Probably related to investigational device
Pain on removing dressing (General disorders) | 1 (1) — Probably related to investigational device
Dressing adhered to the wound/painful (General disorders) | 1 (1) — Possibly related to investigational device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT05873257/Prot_SAP_000.pdf